CLINICAL TRIAL: NCT05959070
Title: Multi-Country Prospective Real-World Study to Validate the CLCI Instrument (DermCLCI-p) in Patients With Moderate-to-Severe Chronic Plaque Psoriasis (IMMagine)
Brief Title: An Observational Study to Validate the Cumulative Life Course Impairment (CLCI) Instrument (DermCLCI-p) in Adult Participants With Moderate to Severe Chronic Plaque Psoriasis (PsO)
Acronym: IMMagine
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-435
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; PsO; Psoriasis; Risankizumab; RZB
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Risankizumab: Participants will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
The IMMagine study aims to validate the newly developed CLCI instrument (DermCLCI-p) in moderate to severe psoriasis (PsO) patients, who will be started on Risankizumb (RZB) treatment and will be enrolled into the validation study up to 28 weeks. The treatment decision for RZB must be made independent of this study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe chronic plaque-type psoriasis diagnosed by a dermatologist and presence of moderate to severe psoriasis symptoms according to physician's clinical judgment at the time of recruitment.
* Participants initiating RZB treatment for psoriasis as per local label. Physician's decision for treatment with risankizumab must have been reached prior to and independently of recruitment in the study.
* Participants able to understand and communicate with the investigator and comply with the requirements of the study.
* Willingness and ability to comply with all study requirements.

Exclusion Criteria:

- Current or recent (within the last 30 days) participation in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult moderate to severe Psoriasis participants treated with labeled dose of Risankizumab.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Validity of the Cumulative Life Course Impairment Instrument (DermCLCI-p) | Baseline through Week 28
  The DermCLCI-p Questionnaire assesses the cumulative impairments in skin diseases. The DermCLCI instrument consists of 30 items and asks participants to consider their disease burden within the last two weeks. Items 1 to 28 are answered on a 4-point Likert scale ranging from 0 (not at all) to 3 (very). Items 29 and 30 are answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very).
Reliability of the Cumulative Life Course Impairment Instrument (DermCLCI-p) | Baseline through Week 28
  The DermCLCI-p Questionnaire assesses the cumulative impairments in skin diseases. The DermCLCI instrument consists of 30 items and asks participants to consider their disease burden within the last two weeks. Items 1 to 28 are answered on a 4-point Likert scale ranging from 0 (not at all) to 3 (very). Items 29 and 30 are answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very).
Responsiveness of the Cumulative Life Course Impairment Instrument (DermCLCI-p) | Baseline through Week 28
  The DermCLCI-p Questionnaire assesses the cumulative impairments in skin diseases. The DermCLCI instrument consists of 30 items and asks participants to consider their disease burden within the last two weeks. Items 1 to 28 are answered on a 4-point Likert scale ranging from 0 (not at all) to 3 (very). Items 29 and 30 are answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (16):
- Belgium (5):
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 252456, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 253234, Brussels, Brussels Capital
  - UZ Gent /ID# 252458, Ghent, Oost-Vlaanderen
  - Dermatologie Maldegem /ID# 252454, Maldegem, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 252457, Leuven, Vlaams-Brabant
- Canada (6):
  - Wiseman Dermatology Research /ID# 255883, Winnipeg, Manitoba
  - Dermatrials Research /ID# 253879, Hamilton, Ontario
  - Lynde Institute for Dermatology /ID# 253876, Markham, Ontario
  - JRB Research /ID# 253877, Ottawa, Ontario
  - SKiN Centre for Dermatology /ID# 255882, Peterborough, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 262591, Saint-Jérôme, Quebec
- Germany (5):
  - Hautarztpraxis Mortazawi /ID# 255872, Remscheid, North Rhine-Westphalia
  - Dermatologische Praxis Dr. med. Marvin Kuske /ID# 265688, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 254340, Hamburg
  - Gemeinschaftspraxis Dres. Anika Hünermund/Mario Pawlak /ID# 255874, Heilbad Heiligenstadt
  - Praxis Dres. Wiemers/Wiemers /ID# 255873, Leipzig

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P23-435